CLINICAL TRIAL: NCT00815750
Title: Decision Making in Unaffected First-Degree Relatives of Prostate Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-15320; 106302 (Other: USF IRB)
Record Dates: First submitted 2008-12-29; First posted 2008-12-30 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase I - Information Gathering (Other)
  Interventions: Other: Information Gathering
- Phase 2 - Decision Aid (Other)
  Interventions: Other: Decision Aid

INTERVENTIONS:
Other: Information Gathering — An information gathering phase leading to development of a new decision aid.
  Arms: Phase I - Information Gathering
Other: Decision Aid — To test the newly developed decision aid.
  Arms: Phase 2 - Decision Aid

SUMMARY:
There are two parts to this study: (1) an information gathering phase leading to development of a new decision aid (phase 1); and (2) a study to test the newly developed decision aid (phase 2).

DETAILED DESCRIPTION:
Phase 1 - The purpose of this part of the research study is to conduct individual interviews and focus groups (group discussions) to learn more about the things or behaviors that help men to stay healthy and the decision making process for prostate cancer screening. We will discuss men's general health concerns, knowledge, beliefs, and concerns regarding prostate cancer and screening for prostate cancer. We will use the results from this study to develop a decision aid to help first-degree relatives of prostate cancer patients make informed decisions about whether to undergo testing or not to undergo testing for prostate cancer. The new decision aid will include a digital videodisc (DVD) and an accompanying booklet. We hope to learn from you the needs and concerns of first-degree relatives, what information to include in the decision aid, what language to use, and the best way to present this information.

Phase 2 - The purpose of this part of the research study is to test the usefulness and acceptability of a new decision aid we developed specifically for first-degree relatives (FDRs) of prostate cancer patients. We will compare the new decision aid to another widely available decision aid that was not developed specifically for first-degree relatives. The goal is to see if the new decision aid will change knowledge (about prostate cancer and screening) and increase satisfaction with decision making (intention or decision made). If we find some evidence that the new decision aid is relevant (useful) and acceptable, we will then do a larger study with several hundred men to determine more definitively whether the new decision aid is better than already existing general decision materials and for which men it works best.

Because the correct decision (whether to undergo screening or not to undergo screening) is not known at this time, the goal of decision aids is to present both (in a balanced manner) the potential harms and benefits of screening. Therefore, this study focuses on the informed decision making (knowledge and satisfaction with decision).

ELIGIBILITY:
Inclusion/Exclusion Criteria:

* Index Patients - African American and White (non-Hispanic) index patients who have completed definitive treatment for prostate cancer will be approached to participate.
* Index Patients Must: (a) reside in the tri-county Tampa Bay area (Hillsborough, Pinellas and Pasco Counties, FL) to simplify logistics of arranging face-to-face focus groups; (b) be willing to attend a focus group; (c) be able to speak, read and write in English; and (d) be able to provide written informed consent.
* Index patients will be asked to nominate at least one male FDR (son or brother) with no history of prostate cancer.
* Unaffected FDRs - Inclusion criteria for FDRs includes: (a) be non-Hispanic African American or White males between the ages of 40 and 70; (b) have no self-reported history of a diagnosis of any form of cancer (excluding non-melanoma skin cancer), (c) have no self-reported history of prostate biopsy, or transrectal ultrasound to investigate or rule out diagnosis of prostate cancer; (d) have not participated in the phase (formative) portion of this study (i.e., must be "naïve" to the intervention); (e) be able to speak, read and write English; (f) self-report access to a DVD player; and (g) be able to provide written informed consent. FDRs with a relative in active definitive prostate cancer treatment (i.e., surgery, radiotherapy or chemotherapy, except for hormone therapy) or who has completed treatment in the past 30 days will not be eligible. FDRs with multiple living relatives who been diagnosed with prostate cancer will be excluded to reduce heterogeneity of our phase 2 sample; this exclusion criterion is expected to have a minimal influence on accrual in light of our previous data on the percentage of men with multiple affected relatives (less than 5%).

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2008-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Aim #1 Formative, Phase 1 | 1 day
  To assess and enhance the Centers for Disease Control and Prevention (CDC)prostate cancer screening decision guides into targeted informed decision aids developed specifically for first-degree relatives of prostate cancer patients.

SECONDARY OUTCOMES:
Aim #2 Pilot Intervention, Phase 2 | 1 year
  To assess the feasibility, acceptability and preliminary efficacy of the enhanced decision aids for first degree relatives of prostate cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Clement Gwede, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (2):
- United States (2):
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - James A. Haley VA Hospital, Tampa, Florida